CLINICAL TRIAL: NCT07097441
Title: Effect of the Use of Atracurium With or Without Reversal Agent on Haemodynamic Parameters During Extubation: a Randomized Controlled Trial
Brief Title: To Observe Haemodynamic Parameters Including, Heart Rate, Blood Pressure, Respiratory Rate , and Oxygen Saturation, With or Without Giving Reversal Agent on Extubation, in Patients Receiving Single Shot of Atracurium , and to Observe Post Operative Residual Paralysis and Airway Reflexes in PACU.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Fariha Ahmed, Resident anaesthesiology R4, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9110824FAANE
Record Dates: First submitted 2025-07-17; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Tachycardia; Hypertension; Hypoxia; Hyperventilation; Residual Paralysis, Post Anesthesia
MeSH Terms: conditions — Tachycardia; Hypertension; Hypoxia; Hyperventilation; Delayed Emergence from Anesthesia | interventions — Saline Solution; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neostigmine group ( Group B ) (Active Comparator): This group will reeive neostigmine ( reversal agent ) at the end of surgery before extubation and then haemodynamic parameters will be observed
  Interventions: Drug: neostigmine (reversal agent)
- normal saline group ( Group A ) (Experimental): This group will receive normal saline ( no reversal ) at the end of surgery before extubation and then haemodynamic parameters will be observed
  Interventions: Drug: Placebo drug ( normal saline )

INTERVENTIONS:
Drug: Placebo drug ( normal saline ) — At the end of surgery patients will be given placebo ( normal saline ) instead of neostigmine ( reversal agent of atracurium ) , to observe Heart rate, blood pressure , respiratory rate and oxygen saturation on extubation and post operative airway reflexes and residual paralysis
  Other Names: Group A
  Arms: normal saline group ( Group A )
Drug: neostigmine (reversal agent) — At the end of surgery patients will be given neostigmine ( reversal agenr ) , to observe Heart rate, blood pressure , respiratory rate and oxygen saturation on extubation and post operative airway reflexes and residual paralysis
  Other Names: Group B
  Arms: Neostigmine group ( Group B )

SUMMARY:
The goal of this clinical trial is to to observe the haemodynamic parameters including Heart Rate Blood pressure Respiratory rate and Oxygen Saturation with or without giving reversal agent on extubation in patients receiving atracurium on induction , it will also observe post operative residual paralysis respiratory depression and airway reflexes in the post anaesthesia care unit Researchers will compare neostigmine which is the reversal agent and the placebo drug by giving it at the end on surgery before extubation to observe haemodynamic parameters The main questions it aims to answer are Will participants have a stable haemodymaics if no reversal ( neostigmine ) is used during extubation Will it provide a safe extubation and no complications post operatively Participants will be given Either neostigmine or placebo drug at the end of surgery before extubation Will be obseved and monitored for two hours postoperatively in the post anaesthesia care unit Will be monitored for post operative complications like respiratory depression or residual paralysis

.

DETAILED DESCRIPTION:
Objective : To observe the haemodynamic parameters including Heart Rate Blood pressure Respiratory rate and Oxygen Saturation with or without giving reversal agent on extubation in patients receiving atracurium on induction , and secondary objective was to observe post operative residual paralysis respiratory depression and cough and gag reflex Study design : Controlled , randomised , and triple Blind trial . Place and duration of study: Dr Ziauddin Hospital Clifton Karachi , from March to June 2025.

Methodology : This was a triple blind study . A total of 100 patients were randomly assigned by the CTU to two groups , the placebo group ( Group A ) and the neoglycopyrolate group (Group B) based on computer generated allocation. At the end of the surgery, patients in Group A were administered IV normal saline and Group B were administered neoglycopyrolate 50 mcg/kg . The primary outcome was to observe heart rate , blood pressure, oxygen saturation and respiratory rate after giving the drug , before extubation , at extubation and at 1mins, 5mins, 10mins, 20mins, and 2h thereafter, while the secondary outcome was to observe post operative airway reflexes and residual paralysis in the post anaesthesia care unit

ELIGIBILITY:
Inclusion Criteria:

* American society of anaesthesiology class 1 and 2
* Surgeries lasting for 60 mins
* .Surgeries requiring general anaesthesia and tracheal intubation and single intubation dose of atracurium

Exclusion Criteria:

* American society of anaesthesiology class 3 and above
* Any previous reaction to atracurium
* Active asthma
* Severe pulmonary cardiac kindney and liver disease

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male and female
Enrollment: 100 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Heart rate | From the time of extubation till discharge from post anaesthesia care unit
  To observe Heart rate, via pulse oximeter and ECG
Blood Pressure | From the time of extubation till discharge from post anaesthesia care unit
  to observe Blood Pressure via Sphygmomanometer
Respiratory Rate | From the time of extubation till discharge from post anaesthesia care unit
  to observe respiratory rate via capnometer
Oxygen Saturation | From the time of extubation till discharge from post anaesthesia care unit
  to observe oxygen saturation via pulse oximeter

SECONDARY OUTCOMES:
Airway reflexes | From the time of extubation till discharge from post anaesthesia care unit
  to observe cough and gag reflex via Binary scale e.g Yes/No
Residual paralysis | From the time of extubation till discharge from post anaesthesia care unit
  to observe head lift for more than 5 secs and firm hand grip via Bonary scale e.g Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Asma Abdus Salam, Consultant anaesthesiology, Study Chair — Ziauddin university clifton
Locations (1):
- Ziauddin university, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berg H, Roed J, Viby-Mogensen J, Mortensen CR, Engbaek J, Skovgaard LT, Krintel JJ. Residual neuromuscular block is a risk factor for postoperative pulmonary complications. A prospective, randomised, and blinded study of postoperative pulmonary complications after atracurium, vecuronium and pancuronium. Acta Anaesthesiol Scand. 1997 Oct;41(9):1095-1103. doi: 10.1111/j.1399-6576.1997.tb04851.x. PMID 9366929
- [Result] Eikermann M, Fassbender P, Malhotra A, Takahashi M, Kubo S, Jordan AS, Gautam S, White DP, Chamberlin NL. Unwarranted administration of acetylcholinesterase inhibitors can impair genioglossus and diaphragm muscle function. Anesthesiology. 2007 Oct;107(4):621-9. doi: 10.1097/01.anes.0000281928.88997.95. PMID 17893459
- [Result] Baillard C, Gehan G, Reboul-Marty J, Larmignat P, Samama CM, Cupa M. Residual curarization in the recovery room after vecuronium. Br J Anaesth. 2000 Mar;84(3):394-5. doi: 10.1093/oxfordjournals.bja.a013445. PMID 10793602
- [Result] Bartkowski RR. Incomplete reversal of pancuronium neuromuscular blockade by neostigmine, pyridostigmine, and edrophonium. Anesth Analg. 1987 Jul;66(7):594-8. PMID 3605668
- [Result] Fragen RJ. Role of reversal agents. J Clin Anesth. 1992 Sep-Oct;4(5 Suppl 1):9S-15S. doi: 10.1016/0952-8180(92)90012-p. No abstract available. PMID 1356374
- [Result] Kirkegaard-Nielsen H, Severinsen IK, Pedersen HS, Lindholm P. Factors predicting atracurium reversal time. Acta Anaesthesiol Scand. 1999 Sep;43(8):834-41. doi: 10.1034/j.1399-6576.1999.430809.x. PMID 10492412
- [Result] Carroll MT, Mirakhur RK, Lowry D, Glover P, Kerr CJ. A comparison of the neuromuscular blocking effects and reversibility of cisatracurium and atracurium. Anaesthesia. 1998 Aug;53(8):744-8. doi: 10.1046/j.1365-2044.1998.00530.x. PMID 9797517
- [Result] 13 .Pollard BJ. Neuromuscular blocking agents and reversal agents. Anaesthesia & intensive care medicine. 2005 Jun 1;6(6):189-92.
- [Result] 12. Nagelhout J, Plaus K. Neuromuscular blocking agents, reversal agents, and their monitoring. Nurse anesthesia. 2017 May 27:179-202.
- [Result] Lee H, Jeong S, Choi C, Jeong H, Lee S, Jeong S. Anesthesiologist's satisfaction using between cisatracurium and rocuronium for the intubation in the anesthesia induced by remifentanil and propofol. Korean J Anesthesiol. 2013 Jan;64(1):34-9. doi: 10.4097/kjae.2013.64.1.34. Epub 2013 Jan 21. PMID 23372884
- [Result] Butterly A, Bittner EA, George E, Sandberg WS, Eikermann M, Schmidt U. Postoperative residual curarization from intermediate-acting neuromuscular blocking agents delays recovery room discharge. Br J Anaesth. 2010 Sep;105(3):304-9. doi: 10.1093/bja/aeq157. Epub 2010 Jun 24. PMID 20576632
- [Result] Reich DL, Mulier J, Viby-Mogensen J, Konstadt SN, van Aken HK, Jensen FS, DePerio M, Buckley SG. Comparison of the cardiovascular effects of cisatracurium and vecuronium in patients with coronary artery disease. Can J Anaesth. 1998 Aug;45(8):794-7. doi: 10.1007/BF03012152. PMID 9793671
- [Result] Use of atracurium and its reversal by anaesthesiologists at a tertiary care hospital. (2013). International Research Journal of Pharmacy, 4(3), 178-181.
- [Result] Babu KC, Rajan S, Sandhya SVK, Raj R, Paul J, Kumar L. Effectiveness and Safety of Extubation before Reversal of Neuromuscular Blockade versus Traditional Technique in Providing Smooth Extubation. Anesth Essays Res. 2021 Jan-Mar;15(1):133-137. doi: 10.4103/aer.aer_78_21. Epub 2021 Aug 30. PMID 34667360
- [Result] Varposhti MR, Heidari SM, Safavi M, Honarmand A, Raeesi S. Postoperative residual block in postanesthesia care unit more than two hours after the administration of a single intubating dose of atracurium. J Res Med Sci. 2011 May;16(5):651-7. PMID 22091288
- [Result] Luo J, Chen S, Min S, Peng L. Reevaluation and update on efficacy and safety of neostigmine for reversal of neuromuscular blockade. Ther Clin Risk Manag. 2018 Dec 10;14:2397-2406. doi: 10.2147/TCRM.S179420. eCollection 2018. PMID 30573962
- [Result] Debaene B, Plaud B, Dilly MP, Donati F. Residual paralysis in the PACU after a single intubating dose of nondepolarizing muscle relaxant with an intermediate duration of action. Anesthesiology. 2003 May;98(5):1042-8. doi: 10.1097/00000542-200305000-00004. PMID 12717123
- [Result] Tsai YH, Chen CY, Wong HF, Chou AH. Comparison of neostigmine and sugammadex for hemodynamic parameters in neurointerventional anesthesia. Front Neurol. 2023 Apr 17;14:1045847. doi: 10.3389/fneur.2023.1045847. eCollection 2023. PMID 37139057
- [Result] Neely GA, Sabir S, Kohli A. Neostigmine. 2025 Jan 19. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470596/ PMID 29261883
- [Result] Hughes R, Chapple DJ. The pharmacology of atracurium: a new competitive neuromuscular blocking agent. Br J Anaesth. 1981 Jan;53(1):31-44. doi: 10.1093/bja/53.1.31. PMID 6161627
- See also: A total of 31 patients were randomized to sugammadex, and 30 patients were randomized to neostigmine. Except for anesthesia time, there were no significant differences in any of the clinical characteristics between the two groups. The results demonstrate — https://www.frontiersin.org/journals/neurology/articles/10.3389/fneur.2023.1045847/full
- See also: orty patients were allocated into two equal groups. In Group E, at the end of surgery, extubation was performed and reversal was administered after extubation. In Group L, reversal was given and patients were extubated in the traditional way. Quality of — https://pubmed.ncbi.nlm.nih.gov/34667360/
- See also: Two hundred and sixteen patients scheduled for elective surgery under general anaesthesia requiring tracheal intubation were included in the study. They received a single intubating dose of intravenous atracurium (0.5 mg/kg) to facilitate tracheal intuba — https://pubmed.ncbi.nlm.nih.gov/22091288/
- See also: the pharmacological properties of atracurium are of sufficient interest to merit its evaluation as a neuromuscular blocking agent in anaesthetized man — https://pubmed.ncbi.nlm.nih.gov/6161627/